CLINICAL TRIAL: NCT00364715
Title: Study the Expression of Annexin A1 and Its Potential Usage as a Prognostic Marker in Oral Cancer
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9561702012
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2006-08-17 (Estimated); Status verified 2006-08

CONDITIONS: Squamous Cell Carcinoma
Keywords: Nuclear localization, annexin A1, oral SCC
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Recent studies have shown that dysregulation of ANXA1 expression are associated with tumorigenesis. Overexpression of ANXA1 protein is found in a wide variety of human tumors, such as breast 10, liver 11, pancreatic cancer14 and glial tumors15. In contrast, reduced levels of ANXA1 protein expression have been reported in ESCC4, 5, gastric6, breast7, head and neck SCC8 and prostate cancer9. No previous study on ANXA1 protein expression has been reported in the cancer of oral cavity. Furthermore, although alterations in annexin expression in different types of tumors have been described, no correlation has been established between ANXA1 and overall patient survival yet.

ANXA1 is a major cellular substrate of the oncogenic tyrosine kinases such as EGF receptor and hepatocyte growth factor (HGF) receptor, c-met. Previously, we have shown that expression of HGF and c-met is significantly associated with the progression of OSCC in Taiwan. Kermorgant et al. recently showed that PKC controls HGF-dependent c-met traffic, signaling and cell migration. Prior study indicate that the mitogen phorbol-12-myristate 13-acetate (PMA) induced ANXA1 nuclear translocation in a PKCdelta-dependent manner and ANXA1 nuclear translocation may participate in the regulation of cellular proliferation and the differentiation. However, it is not known whether HGF can induce ANXA1 nuclear translocation or not and how this relates to the pathogenesis of oral SCC.

In this study we aimed to investigate whether HGF induced the translocation of ANXA1 protein to the nucleus in OSCC cells and the role(s) of ANXA1 nuclear localization in the carcinogenesis of OSCC using an immunohistochemical technique. The data suggest a novel mechanism for HGF-induced ANXA1 protein nuclear translocation that may play an important role in the pathogenesis and prognosis in oral SCCs.

DETAILED DESCRIPTION:
MATERIAL AND METHODS

After approval by the Hospital Review Board, we obtained formalin-fixed, paraffin-embedded specimens from 115 patients with primary oral SCC and 66 patients with oral ED at the Department of Pathology, National Taiwan University Hospital, Taipei, Taiwan. Diagnosis of oral SCC and ED was based on histological examination of hematoxylin and eosin-stained tissue sections. All patients received total surgical excision of the lesions at the Department of Oral and Maxillofacial Surgery or Department of Otolaryngology, National Taiwan University Hospital during the period from 1997 to 2004. Specimens were obtained from either incisional biopsies or total surgical excision of the lesions. If lymph node was diagnosed as positive for SCC, neck dissection and postoperative radiation therapy were also included in the treatment protocol. No patient had received any cancer therapy before initial biopsies. Details of the patients' oral habits, including daily consumption of AQs, cigarettes, and alcohol as well as the duration of these habits, were also recorded in the medical chart. Twenty biopsy specimens of normal oral mucosa (NOM) were obtained from non-AQ-chewers and non-smokers during extraction of impacted permanent lower third molars after obtaining informed consent, and used as the healthy controls.

Cell culture Dulbecco's modifed Eagle's medium (DMEM), and fetal bovine serum (FBS) were purchased from Life Technologies, Inc. (Gaithersburg, MD,USA). PD98059, Ly294002, SB203580 and Hepatocyte growth factor (HGF) were products of Sigma (St Louis, MO, USA). Anti-ANX-1 monoclonal antibody was purchased from BD Biosciences (Lexington, KY, USA). Cell culture SAS cells were maintained in DMEM supplemented with 10% heat-inactivated FBS, penicillin (100 UAmL)1), and streptomycin (100 lgAmL)1) at 37 o C under 5% CO2 atmosphere. For Western blot analysis, cells were seeded into 10 cm dishes at 2 x 106 cells per dish. After 18-24 hr, cells were further grown in the same medium supplemented without FBS for 24 h. Serum-starved cells were treated with HGF in the indicated times. For immunostaining, 2 x 105 cells grown on cover slides (22 x 22 mm) were starved for 24 h before stimulation with HGF.

Pre-treatment with PD098059, Ly294002 and SB203580 The cells were plated overnight in complete medium and then washed. The cells cultured in serum-free DMEM were pre-treated with 50M PD098059 (inhibitor of ERK), 30 M Ly294002( inhibitor of PI-3 kinase) and 20 M SB203580(inhibitor of p38) for 3 hrs respectively, and then they were treated with 40ng HGF for 3hrs. The cells were checked by immunohistochemistry and Western blot with ANXA1 antibody.

Immunocytochemistry(IHC) Formalin-fixed, paraffin-embedded tumor samples were assessed for annexin A1 expression.The IHC procedures was followed as the reference18, The monoclonal primary antibody anti-Annexin AI(1:600 dilution), directed against the the N-terminus of annexin 1 were obtained from a signal source (BD Biosciences). Protein translocation as determined by two pathologists (Jeng and Lin) using immunohistochemistry was scored as negative (score 0), positive (score 1) and cytoplasmic protein expression was scored as negative (score 0), weak (score 1), moderate (score 2), or strong (score 3) using a system that has been previously validated.

SAS cells grown on cover slides were fixed with 3.7% paraformaldehyde for 15 min and permeabilized with 0.2% Triton X-100 in PBS (0.58M Na2HPO4, 0.17 M Na H2PO4, 0.68 M NaCl, pH=7.4)(PBST) for 5 min. After washing the cells with PBST three times, the cells were blocked for 30 min in PBS containing 1% bovine serum albumin. Immunostaining was performed by incubation with anti-ANX-1 monoclonal antibody (1:800 dilution) for 2h. After washing the cells with PBST three times, the cells were incubated with TRITC-conjugated rabbit anti-(mouse IgG) Ig for 1 h. Cover slides were washed with PBST, mounted, and examined using a Leica TCS SP2 Confocal microscope (Leica Microsystems, Wetzlar GmBH, Germany).

Cell fractionation SAS cells were seeded into 10cm dishes at 2x 106 cells/dish and cultured in DMEM for 18-24 h. The cells were starved for 24 h in serum-free media. After treatment with HGF for a given time, the cells were harvested and washed with ice-cold PBS. The cells were then resuspended in 100 lL of lysis buffer (10 mM Hepes, 10 mM NaCl, 0.1 mM EDTA, 0.1 mM EGTA, 1% NP-40, 0.5 mM phenylmethylsulfonyl uoride, 0.1 mM dithiothreitol, 0.1 mM sodium orthovanadate, and protease inhibitors) and incubated on ice for 10 min. The nuclei were collected by centrifugation at 2000 g for 5 min at 4 o C. The supernatant was collected as a cytosolic fraction. Protein concentration of each sample was determined.

Evalution of annexin A1 Protein Expression The distributions of ANXA1 expression in four categories (0-25%, 26-50%, 51-75% and 76-100%) with nuclear translocation were firstly showed by clinicopathological parameters of the oral ED and SCCs and the correlations between mean levels of expression and these clinicopathological parameters were further examined using ANOVA. The Kaplan-Meier product-limit method was used to assess the prognostic significance of the ANXA1 nuclear staining in cancer cells as well as other clinicopathological parameters. Comparison of cumulative survival between groups was performed using the log-rank test with the Statistica program (StatSoft Inc., USA). Multivariable analyses were performed with Cox regression model to assess additional prognostic values of the different variables using SAS 8.0 (SAS Institute Inc., USA). A P-value of less than 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

noraml, dysplasia, SCC

Exclusion Criteria:

Ages: 26 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Mark YP Kuo, PHD, Principal Investigator — National Taiwan University , Dental Department
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/